CLINICAL TRIAL: NCT05539586
Title: Effectiveness of Tecar Therapy in Patients With Chronic Achilles Tendinopathy. Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Tecar Therapy in Patients With Chronic Achilles Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Maxim Canet Vintró, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBSCFCTEC
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Achilles Tendinopathy
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tecar group (Experimental)
  Interventions: Other: Tecartherapy
- Sham Group (Sham Comparator)
  Interventions: Other: Sham

INTERVENTIONS:
Other: Tecartherapy — Patients will receive therapeutic exercise sessions for 7 weeks and 7 tecartherapy sessions.
  Arms: Tecar group
Other: Sham — Patients will receive therapeutic exercise sessions for 7 weeks and 7 sessions of simulated tecartherapy.
  Arms: Sham Group

SUMMARY:
Achilles tendinopathy is characterized by pain, decreased performance and swelling in and around the tendon. Up to 29% of patients with Achilles tendinopathy may require surgical intervention. It can be complicated by partial tears or complete rupture, placing a long-term burden on the healthcare system and making treatment more difficult.

The most common location of Achilles tendinopathy is in the insertional area of the calcaneus, 1.5 to 2 cm cranial to the bone. The most common location of pathologic inflammation was at the fascial intersection of the medial gastrocnemius and soleus when fused with the proximal Achilles tendon (66% of patients and the distal part of the Achilles tendon near the calcaneus. The four cornerstones of tendon histopathology are: cellular activation and increased cell number, increased ground substance, collagen disorganization and neovascularization. In addition, blood supply is one of the most influential factors in tendon tissue repair. A recent clinical trial compared the outcome after low frequency microwave hyperthermia with traditional ultrasound. The hyperthermia group recorded significantly better results after treatment and one month later. The use of deep heating modalities, due to their beneficial effects of increased circulation and cellular metabolism resulting in increased waste and nutrient exchange in a specific area, has long been accepted as part of the treatment of overuse tendinopathies . The application of heat has been reported to improve blood flow and oxygen saturation in the Achilles tendon.Physical therapies based on electrical or electromagnetic stimulation have been used in rehabilitation, in some cases combining electrical therapy with radiofrequency. Specifically, resistive capacitive electrical transfer therapy (CRet) has been used in physical rehabilitation and sports medicine to treat muscle, bone, ligament and tendon injuries. CRet is a non-invasive electrothermal therapy classified as deep thermotherapy, which is based on the application of electrical currents within the radiofrequency range of 300 kHz - 1.2 MHz. he effects attributed to this technique include increased deep and superficial blood circulation, vasodilatation, increased temperature, elimination of excess fluid and increased cell proliferation. Some of these reactions, such as increased blood perfusion, are known to be related to the increase in temperature, but others, such as increased cell proliferation, appear to be primarily related to the passage of current. There are currently numerous treatment proposals for this pathology, however, the only one that has shown significant improvements are eccentric exercise protocols. The only drawback of this type of exercise is that the results are obtained in the long term.

There is currently no study that has compared the effectiveness of adding a tecartherapy protocol to the eccentric exercise protocol in chronic Achilles tendinopathy in athletes in the short and medium term in both functional and structural variables.

DETAILED DESCRIPTION:
Achilles tendinopathy is characterized by pain, decreased performance and swelling in and around the tendon. Up to 29% of patients with Achilles tendinopathy may require surgical intervention. It can be complicated by partial tears or complete rupture, placing a long-term burden on the healthcare system and making treatment more difficult.

The most common location of Achilles tendinopathy is in the insertional area of the calcaneus, 1.5 to 2 cm cranial to the bone. The most common location of pathologic inflammation was at the fascial intersection of the medial gastrocnemius and soleus when fused with the proximal Achilles tendon (66% of patients and the distal part of the Achilles tendon near the calcaneus. The four cornerstones of tendon histopathology are: cellular activation and increased cell number, increased ground substance, collagen disorganization and neovascularization. In addition, blood supply is one of the most influential factors in tendon tissue repair. There is an animal study in which when the blood supply to the Achilles tendon of a rabbit was decreased, the following changes were observed: the normally attached fascicles of the rabbit tendon separated and the tenocytes became disorganized from the interfascicular spaces. Collagen filaments became acellular and fragmented. Furthermore, it was shown that the changes observed in chronic degenerative tendon disorders in humans are the same as those that occur when the blood supply to the rabbit Achilles tendon is disturbed. This demonstrates that vascular supply is one of the important factors in treating tendon tissue.

A recent clinical trial compared the outcome after low frequency microwave hyperthermia with traditional ultrasound. The hyperthermia group recorded significantly better results after treatment and one month later. The use of deep heating modalities, due to their beneficial effects of increased circulation and cellular metabolism resulting in increased waste and nutrient exchange in a specific area, has long been accepted as part of the treatment of overuse tendinopathies . The application of heat has been reported to improve blood flow and oxygen saturation in the Achilles tendon. Thus, thermal agents may be an effective method to treat this type of tendon disorders.

Physical therapies based on electrical or electromagnetic stimulation have been used in rehabilitation, in some cases combining electrical therapy with radiofrequency. Specifically, resistive capacitive electrical transfer therapy (CRet) has been used in physical rehabilitation and sports medicine to treat muscle, bone, ligament and tendon injuries. CRet is a non-invasive electrothermal therapy classified as deep thermotherapy, which is based on the application of electrical currents within the radiofrequency range of 300 kHz - 1.2 MHz. While the heat conducted by surface thermotherapy cannot reach the muscle due to the electrical resistance of the tissues, the capacitive-resistive electric currents in CRet therapy can generate heating of deep muscle tissues, which in turn improves hemoglobin saturation. In Europe, CRet is widely used in various medical rehabilitation processes. The physiological effects of this type of physiotherapy are generated by the application to the human body of an electromagnetic field with a frequency of approximately 0.5 MHz. The effects attributed to this technique include increased deep and superficial blood circulation, vasodilatation, increased temperature, elimination of excess fluid and increased cell proliferation.

Some of these reactions, such as increased blood perfusion, are known to be related to the increase in temperature, but others, such as increased cell proliferation, appear to be primarily related to the passage of current.

It is also true that this increase in tissue temperature, generated through the application of the device, is a physical reaction to the passage of the current (Joule effect). Although there are already clinical publications that support this mechanism, the amount of energy and current that must be transferred to obtain the desired temperature increase is unknown. Moreover, the control of these reactions, by adjusting parameters such as absorbed power and electrode position, are still largely based on the empirical experience of therapists.

Recently, new cadaveric publications have been published that support the mechanisms of current flow and thermal changes in this situation, especially a study by López-de-Celis et al. in which the thermal effects and current flow in the myotendinous junction of the medial gastrocnemius and Achilles tendon were demonstrated.

With this background, in which thermal effects, current passage and symptomatic improvements have been demonstrated in patients with pathology, the possibility that these treatments improve functional sports capabilities is raised. This hypothesis arises from the fact that the passage of current and thermal changes have been directly related to viscoelastic changes in capsular and muscular tissue. There are currently numerous treatment proposals for this pathology, however, the only one that has shown significant improvements are eccentric exercise protocols. The only drawback of this type of exercise is that the results are obtained in the long term.

There is currently no study that has compared the effectiveness of adding a tecartherapy protocol to the eccentric exercise protocol in chronic Achilles tendinopathy in athletes in the short and medium term in both functional and structural variables.

Recently, new cadaveric publications have been published that support the mechanisms of current flow and thermal changes in this situation, especially a study by López-de-Celis et al. in which the thermal effects and current flow in the myotendinous junction of the medial gastrocnemius and Achilles tendon were demonstrated.

With this background, in which thermal effects, current passage and symptomatic improvements have been demonstrated in patients with pathology, the possibility that these treatments improve functional sports capabilities is raised. This hypothesis arises from the fact that the passage of current and thermal changes have been directly related to viscoelastic changes in capsular and muscular tissue. There are currently numerous treatment proposals for this pathology, however, the only one that has shown significant improvements are eccentric exercise protocols. The only drawback of this type of exercise is that the results are obtained in the long term.

There is currently no study that has compared the effectiveness of adding a tecartherapy protocol to the eccentric exercise protocol in chronic Achilles tendinopathy in athletes in the short and medium term in both functional and structural variables.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must have signed the informed consent form in order to evaluate their participation in the study.
* Actively practice some sporting activity.
* Have a medical diagnosis of chronic Achilles tendinopathy of more than 3 months of evolution.
* Not having previously received any tecartherapy treatment.
* Be over 18 years of age.

Exclusion Criteria:

* Volunteers who have suffered a sports injury during the last two months or are unable to perform physical activity.
* Subjects with bilateral tendinopathies.
* Subjects who report allergies to the conductive cream.
* Not understanding the information provided by the therapist.
* Participating in other research studies.
* Subjects undergoing pharmacological medical treatment that may interfere with the measurements, such as treatment with anticonvulsants, antidepressants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in numerical pain rating scale (0-10) | Baseline; 3 weeks follow-up; 7 weeks follow-up
  EVA pain scale will be used, where the patient will tell us the pain in numerical form.
Change in visual analogue scale (0-100 mm) | Baseline; 3 weeks follow-up; 7 weeks follow-up
  EVA pain scale will be used, where the patient will point on a fingertip on a straight line without numbers which has been his perception of pain.

SECONDARY OUTCOMES:
Strength (kilograms) | Baseline; 3 weeks follow-up; 7 weeks follow-up
  To measure the strength of the gastrocnemius muscles, a precision dynamometer (Microfeet II) will be used and the maximum force will be analyzed during an isometric contraction of this musculature for 5 seconds. The participant will be placed in supine decubitus with his ankle close to a wall. The dynamometer (Microfeet II) will be placed between the foot and the wall at the level of the metatarsals. The participant will be asked to perform a maximum plantar flexion for five seconds against the dynamometer. The maximum force in kilograms performed by the subject during this test will be recorded.
Ankle range of motion in loading (degrees) | Baseline; 3 weeks follow-up; 7 weeks follow-up
  The measurement of ankle dorsal flexion range of motion in loading is a variable to be studied. A universal goniometer will be used. The patient will lean against a wall and keeping the heel on the floor will perform the maximum possible dorsal ankle flexion under load until the first sensation of tension. The goniometer will be aligned with one limb parallel to the ground and the other in the direction of the tibia.
VISA-A questionnaire | Baseline; 3 weeks follow-up; 7 weeks follow-up
  Victorian Institute of Sport Assessment-Achilles Questionnaire, 0-100, higher scores mean a better outcome.
GROC scale | Baseline; 3 weeks follow-up; 7 weeks follow-up
  Global Rating of Change Scale, (-7) - (+7), higher scores mean a better outcome.
Cross-sectional area (mm2) | Baseline; 3 weeks follow-up; 7 weeks follow-up
  The cross-sectional section will be measured using a tracing ellipse method with the trace at the edge of the echogenic bony region. The tendon structure will be evaluated and interpreted as abnormal if there are persistent variations in the homogeneous structure, including a hypoechoic signal, hyperechoic signal, peritendinous fluid collection, contour defect or focal thickening of the tendon and noted. In addition, the images will be evaluated by a grayscale detection program capable of detecting intra-tendon changes imperceptible to the human eye.
Stinfess (N m -1 ) | Baseline; 3 weeks follow-up; 7 weeks follow-up
  Measured by myotonometry. It is determined by the relation between the force produced by the mechanical impulse and the depth of tissue deformation.
  Stiffness should be measured at the point where the patient reports the most pain.
Longitudinal section (mm) | Baseline; 3 weeks follow-up; 7 weeks follow-up
  Thickness will be measured at the point with the largest anteroposterior diameter.